CLINICAL TRIAL: NCT00987298
Title: Technical Validation of Lunar iDXA (GE Healthcare) Visceral Fat Tool
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sanjiv Kaul, M.D. / Head, Division of Cardiovascular Medicine, Oregon Health & Science University / Division of Cardiovascular Medicine
Other Study IDs: OHSU-090320
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Obesity
Keywords: Abdominal Fat; Visceral Fat; Subcutaneous Fat; Dual-energy x-ray absorptiometry; DXA; Computed Tomography; CT; Body Mass Index; Body composition; Percent fat; Waist circumference; Hip circumference
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Visceral fat mass: The study population will include adult men and women, ages 18 to 90 years. All subjects will be recruited at Oregon Health and Science University (OHSU). Subjects will represent a wide range of BMI values (18.5 - 40 kg/m2).
  Interventions: Device: Visceral fat mass measurement

INTERVENTIONS:
Device: Visceral fat mass measurement — Total body DXA measurement, Abdominal CT scan
  Other Names: Lunar iDXA (GE Healthcare)

SUMMARY:
The goal of this project is to compare visceral fat measurements derived from Lunar iDXA total body scans and from Computed Tomography (CT) scans of the abdominal region.

DETAILED DESCRIPTION:
Obesity is one of the greatest public health challenges of the 21st century. The World Health Organization (WHO) estimates for 2005 indicate approximately 1.6 billion adults are overweight (body mass index (BMI) > 25 kg/m2), with 400 million being characterized as obese (BMI > 30 kg/m2). By 2015, the WHO projections predict that the populations of overweight and obese adults will increase to 2.3 billion and 700 million respectively. The major determinant of obesity is the energy imbalance between calorie intakes and expenditures, which can be ascribed to a global dietary shift in favor of energy-dense foods particularly rich in fat and carbohydrates, and a global trend towards sedentary behaviors.

Body fat distribution and abdominal fat in particular is correlated with increased risk of cardiovascular disease, diabetes, hypertension, nonalcoholic fatty liver disease, cancer, and total mortality. It is therefore important to develop minimally invasive clinical tools to assess visceral fat. Computed Tomography (CT) and Magnetic Resonance Imaging (MRI) represent the gold standards for the quantification of visceral and abdominal fat. However, the analytical cost and the limited availability of these instruments for large-scale screenings have encouraged the development of alternative methods based on cost effective and widely distributed technologies. Dual-energy x-ray absorptiometry (DXA) is a promising technology to fill this gap. DXA is being used increasingly as a rapid, precise, and accurate method for measurement of regional and total body composition in both clinical and research settings. Total body assessment using DXA provides a unique capability of non-invasive measurement of skeletal bone status, as well as lean and fat tissue components including percent fat, lean tissue mass, and the android (waist)/gynoid (hip) fat ratio. The DXA technology is well suited to large-scale screening for assessing body composition and fat distribution as a part of a global assessment of metabolic status.

A recent study of a cross-sectional sample of 5440 US adults participating in the NHANES surveys 1999-2004 showed that 29.2% of obese men and 35.4% of obese women (a total of approximately 19.5 million US adults) are metabolically healthy, (sometimes referred to as "uncomplicated" obesity), whereas 30.1% of normal-weight men and 21.1% of normal-weight women (a total of approximately 16.3 million US adults) exhibit clustering of two or more cardiometabolic abnormalities. This study concluded that additional research is required to understand the physiological mechanisms underlying these differences. Another recent study of more than 3000 participants drawn from the Framingham Heart Study showed that both subcutaneous fat and visceral fat were correlated with metabolic risk factors. However, only the effects of visceral fat remain significant after adjusting for common anthropometric indices such as waist circumference and BMI. The issues surrounding cardiometabolic risk among different phenotypes along with the increased risks associated with visceral fat suggests the need to measure visceral adipose tissue in a diverse population.The gold standard, CT, is not a practical solution due to the cost and radiation exposure associated with the measurement. Therefore, it is important to develop a low-cost, low-radiation screening method for measuring visceral adipose tissue.

The present study aims at measuring abdominal fat distribution (CT scan and Lunar iDXA) in 120 adults. These data provide the possibility to validate a new method for measuring abdominal fat distribution (visceral versus subcutaneous fat) against the gold standard, CT. If validated, such a protocol based on Lunar iDXA could offer a rapid and cost effective diagnostic tool for fat distribution assessment of individuals as a basis for future personalized and health care programs.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 90
* BMI: 18.5 - 40
* Subject willing to provide informed consent

Exclusion Criteria:

* Subject who is affected by any diagnosed eating disorder
* Pregnancy
* Subject who is unable or unwilling to give consent
* Subjects who may not be good trial participants based on investigator's discretion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age between 18 and 90 BMI between 18.5 and 40
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Agreement between Lunar iDXA and CT measured visceral fat of the abdominal region | At the time of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Kaul, MD, Principal Investigator — Oregon Health and Science University; David Ergun, PhD, Study Director — GE Healthcare Lunar
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States